CLINICAL TRIAL: NCT02317107
Title: A Longitudinal Examination of Dynamic Balance Control, Vestibular/Ocular Motor Function, and Activity Participation Following Concussion
Brief Title: Examination of Balance, Vestibular, and Ocular Functions and Activity Following Concussion
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, David R Howell, Research Fellow, Boston Children's Hospital
Other Study IDs: IRB-P00016317
Record Dates: First submitted 2014-12-11; First posted 2014-12-15 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Brain Concussion
Keywords: Gait; Mild Traumatic Brain Injury; Post-Concussion Syndrome; Recovery of Function; Locomotion; Motor Activity
MeSH Terms: conditions — Brain Concussion; Post-Concussion Syndrome; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Concussion: Individuals who report to the Division of Sports Medicine at Boston Children's Hospital will be identified for inclusion in the study if they receive a diagnosis of concussion, defined as a complex pathophysiological process affecting the brain, induced by biomechanical forces. If they agree to participate, they will be placed in the concussion group and assessed at each visit to the clinic. No intervention will be administered.
- Control: Individuals who report to the Division of Sports Medicine at Boston Children's Hospital will be identified for inclusion in the study if they come to the clinic for an injury unrelated to brain function or a lower extremity function (which may affect normal gait patterns). If they agree to participate, they will be placed in the control group and assessed at each visit to the clinic. No intervention will be administered.

SUMMARY:
Previous research and position statements have outlined the necessity of balance and gait testing in the post-concussion evaluation of athletes. However, many of the currently available balance testing techniques lack objectivity and sensitivity to the effects of concussion. Such balance impairments may exist following concussion due to disruption of vestibular and/or ocular motor systems. However, no clinically feasible tools have been longitudinally examined to detect gait balance control deficits or to investigate how vestibular or motor dysfunction may lead to gait imbalance. Additionally, participation in physical and cognitive activities post-concussion may affect recovery. While limited evidence exists to support this notion, further investigation is necessary to improve clinical management recommendations.

The proposed study will allow for the examination of tools which add value to post-concussion clinical evaluations and study-related outcomes will enhance the understanding of dynamic balance control and vestibular/ocular motor recovery, and their potential for implementation into concussion management protocols.

DETAILED DESCRIPTION:
To address study hypotheses, the investigators plan to recruit subjects who have been diagnosed with a concussion by participating sports medicine physicians at the Boston Children's Hospital Sports Concussion Clinic. If patients elect to participate, they will undergo their regularly scheduled clinical examination along with two testing components requiring less than 15 minutes of additional time to complete: an instrumented gait balance assessment, a vestibular-ocular motor screen, and a weekly activity survey. Participants with concussion will be matched with control subjects who meet similar demographic characteristics and report to the clinic for other orthopedic injuries that do not affect brain function, gait, or either lower extremity.

During the assessment, participants will complete a protocol which measures balance control while walking and simultaneously completing a cognitive task, a vestibular-ocular motor ability, and physical and cognitive activity levels. As a need exists to develop protocols which utilize inexpensive, objective, and sensitive measurements to track concussion recovery, this study seeks to incorporate innovative and clinically feasible methods into the clinical examination of concussion.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 12 and 40 years
2. No history of concussion in the past year, and no lifetime history of more than 3 concussions
3. Diagnosed with concussion within the past 21 days (concussion group only)

Exclusion Criteria:

1. Lower extremity deficiency or injury, which may affect normal balance or gait
2. History of permanent memory loss
3. Diagnosis of Attention Deficit Disorder (ADD), Attention Deficit Hyperactivity Disorder (ADHD), learning disability, Down syndrome, or developmental delay

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients will come from Boston Children's Hospital and The Micheli Center for Sports Injury Prevention. Concussion will be defined consistent with the latest best-practice consensus statement on concussion in sport as a brain injury defined as a complex pathophysiological process affecting the brain, induced by biomechanical forces. Informed consent will be obtained after study explanation and sufficient time to answer all study-related questions at each respective location.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2015-06-30 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Dynamic Balance Control | 1 year
  For balance control measures, the primary data will come from accelerometers placed on specific anatomical landmarks to assess whole body movement. Peak accelerations and velocities of an estimated center-of-mass during gait under single-task and dual-task conditions will identify how divided attention tasks affect whole body balance control.

SECONDARY OUTCOMES:
Temporal/Distance Gait Measurements | 1 year
  Stride velocity, stride length, gait cycle time, turning duration/velocity, and anticipatory postural adjustments will help to quantify gait stability in different conditions
Vestibular-Ocular Motor Screen | 1 year
  The severity of symptom provocation in each condition of the vestibular-ocular motor test
Weekly physical and cognitive activity scores | 1 year
  Scores rated by the patient will be calculated across their duration of participation in the study and used to associate the amount of activity participated in with the duration of time to recovery

CONTACTS AND LOCATIONS:
Overall Officials: William P Meehan III, MD, Study Chair — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Howell DR, O'Brien MJ, Raghuram A, Shah AS, Meehan WP 3rd. Near Point of Convergence and Gait Deficits in Adolescents After Sport-Related Concussion. Clin J Sport Med. 2018 May;28(3):262-267. doi: 10.1097/JSM.0000000000000439. PMID 28742610
- [Background] Howell DR, Stracciolini A, Geminiani E, Meehan WP 3rd. Dual-task gait differences in female and male adolescents following sport-related concussion. Gait Posture. 2017 May;54:284-289. doi: 10.1016/j.gaitpost.2017.03.034. Epub 2017 Apr 1. PMID 28384609
- [Background] Howell DR, Beasley M, Vopat L, Meehan WP 3rd. The Effect of Prior Concussion History on Dual-Task Gait following a Concussion. J Neurotrauma. 2017 Feb 15;34(4):838-844. doi: 10.1089/neu.2016.4609. Epub 2016 Sep 14. PMID 27541061
- [Background] Howell DR, Brilliant A, Berkstresser B, Wang F, Fraser J, Meehan WP 3rd. The Association between Dual-Task Gait after Concussion and Prolonged Symptom Duration. J Neurotrauma. 2017 Dec 1;34(23):3288-3294. doi: 10.1089/neu.2017.5191. Epub 2017 Oct 16. PMID 28895490
- [Background] Berkner J, Meehan WP 3rd, Master CL, Howell DR. Gait and Quiet-Stance Performance Among Adolescents After Concussion-Symptom Resolution. J Athl Train. 2017 Dec;52(12):1089-1095. doi: 10.4085/1062-6050-52.11.23. Epub 2017 Nov 20. PMID 29154694